CLINICAL TRIAL: NCT02821793
Title: Expectations and Priorities of Elderly Patients for a First Medical Treatment for Cancer : PRIORITY Study
Brief Title: Expectations and Priorities of Elderly Patients for a First Medical Treatment for Cancer
Acronym: PRIORITY
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Fondation Université de Bordeaux (Unknown); AG2R La Mondiale (Other)
Responsible Party: Sponsor
Other Study IDs: IB 2015-06
Record Dates: First submitted 2016-06-14; First posted 2016-07-04 (Estimated); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Kidney Cancer; Lung Cancer; Prostate Cancer; Sarcoma; Ovarian Cancer; Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Kidney Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Sarcoma; Ovarian Neoplasms; Lymphoma | interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elderly patient (70 years and older)
  Interventions: Other: Geriatric consultation, evaluation questionnaire
- Young patient (18 years - 69 years)
  Interventions: Other: Consultation, evaluation questionnaire

INTERVENTIONS:
Other: Consultation, evaluation questionnaire — Consultation, evaluation questionnaire
  Groups: Young patient (18 years - 69 years)
Other: Geriatric consultation, evaluation questionnaire — Geriatric consultation, evaluation questionnaire
  Groups: Elderly patient (70 years and older)

SUMMARY:
The main objective of study is to describe the priorities of elderly patients (70 years and over) undergoing a first medical treatment for cancer, at initiation of treatment and after 3 months of treatment. The main criterion is a prioritization of 4 items per patient from a list of 8 expectations regarding the objectives of their treatment: treatment efficacy, life expectancy, autonomy, daily activities, social activities, heaviness of treatment, toxicity, economics.

DETAILED DESCRIPTION:
For the primary endpoint assessment, this self-administered patient questionnaire will used an opinion scale (Not at all, A little, Moderately, Enough, Many) to explore the eight domains. Next to the completion of the expectations questionnaire, patients will have to order 4 of the different 8 items that they prioritized in regard of the first line treatment that has just been prescribed by their physician.

Secondary endpoint will focus on those 8 proposed expectations of patients at different periods of time since treatment initiation. Patients' priorities will be compared to physician's priorities (using the same prioritization grid) before medical treatment and after 3 months of treatment and to younger patients' priorities (18-69 years). Associations between elderly patients' characteristics (social, medical…) and their priorities will be search.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female:

   1. Age ≥ 70 years
   2. Aged 18-69 years (case population)
2. ECOG / performance status 0-3 (WHO).
3. First line of medical oncology treatment (chemotherapy, targeted therapy, hormone therapy, combination):

   1. Neo-adjuvant setting,
   2. Adjuvant setting: previous neo-adjuvant treatment is allowed,
   3. Metastatic setting: previous neo-adjuvant and/or adjuvant treatment are allowed,
4. Solid tumors (breast, colorectal, kidney, lung, prostate, sarcoma, and ovarian) and lymphoma (indolent and aggressive).
5. Life expectancy of more than 3 months.
6. Patients potentially compliant with the rules of the follow-up study.
7. Patients affiliated to a social security scheme.
8. Patients who received clear information from the investigator on the study and had not refused to participate.

Exclusion Criteria:

1. Exclusive surgery treatment.
2. Exclusive radiotherapy treatment or in combination with oncological medical treatment (concomitant radio-chemotherapy or radio-hormonotherapy).
3. Previous first line of oncological medical treatment in the same indication as the one concerned by the inclusion:

   1. Neo-adjuvant setting: previous line(s) of neo-adjuvant medical treatment,
   2. Adjuvant setting: previous line(s) of adjuvant medical treatment,
   3. Metastatic setting: previous line(s) of metastatic medical treatment,
4. Supportive care without specific medical treatment
5. Previous or ongoing cancer under treatment at the time of inclusion.
6. Patient already included in this study
7. Patient who for psychological, psychiatric, social, family or geographical reasons could not be regularly monitored according to the criteria of the study; patient private of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 patients aged 70 years old or more and 100 patient between 18 and 69 years old.
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2016-01; Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from January 2016 to January 2022 in 8 centers.
Pre-assignment Details: Elderly patients (≥ 70 years of age) were recruited by the investigating oncologists or geriatricians at organ-specific multidisciplinary consultation meetings (RCP) or during consultations.
  Younger patients were identified and recruited in the same way, mainly through RCP or specialized consultation by oncologists.
Period: Overall Study
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Started | 246 | 100
Major Deviation From Protocol | 13 | 0
Major Deviation on Eligibility Criteria | 6 | 1
Completed | 227 | 99
Not Completed | 19 | 1

BASELINE CHARACTERISTICS:
Population: Eligible population : Patients without major deviation on study protocol and eligibility criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years) | Total
Number analyzed (Participants) | 227 | 99 | 326
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 79.2 [75.4 to 96.6] | 61.3 [54.2 to 66.4] | 75.9 [67.7 to 96.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 71 | 220
  Male | 78 | 28 | 106
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 227 | 99 | 326

OUTCOME MEASURES:

1. Primary Outcome: Priorities of Patients Receiving First Medical Treatment for Cancer at Treatment Initiation
Description: Prioritization among of the 4 items selected from a list of 8 expectations regarding the objectives of their treatment : treatment efficacy, life expectancy, autonomy, daily tasks, social activities, burden of treatment, toxicity and economic burden.
  For each expectation, the number and rate of priorization are reported.
Time Frame: Day 0 initiation of treatment
Population: Patients without major deviation on study protocol and eligibility criteria who indicated at least one priority in the prioritization grid at the initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Number analyzed (Participants) | 211 | 97
Participants
  Treatment efficacy | 199 | 93
  Life expectancy | 141 | 80
  Autonomy | 181 | 67
  Daily tasks | 115 | 44
  Social activities | 80 | 47
  Burden of treatment | 47 | 17
  Toxicity | 66 | 35
  Economic burden | 13 | 5

2. Primary Outcome: Priorities of Patients Receiving First Medical Treatment for Cancer 3 Months After Initiation of Treatment
Description: as for outcome 1
Time Frame: 3 months after initiation of treatment
Population: Patients without major deviation on study protocol and eligibility criteria who indicated at least one priority in the prioritization grid 3 months after initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Number analyzed (Participants) | 155 | 88
Participants
  Treatment efficacy | 145 | 85
  Life expectancy | 105 | 72
  Autonomy | 134 | 66
  Daily tasks | 93 | 44
  Social activities | 69 | 46
  Burden of treatment | 27 | 8
  Toxicity | 30 | 22
  Economic burden | 15 | 7

3. Secondary Outcome: Expectations of Patients at Initiation of Treatment
Description: Patients had to rate on a 5-point Likert scale (not at all / a little / moderately / quite / a lot) their expectations for treatment efficacy, life expectancy, autonomy, daily tasks, social activities, burden of treatment, toxicity and economic burden
Time Frame: Day 0 initiation of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Number analyzed (Participants) | 211 | 97
Participants
  Treatment efficacy: Not at all | 3 | 0
  Treatment efficacy: A little | 4 | 0
  Treatment efficacy: Moderately | 5 | 0
  Treatment efficacy: Quite | 24 | 4
  Treatment efficacy: A lot | 173 | 91
  Treatment efficacy: Missing | 2 | 2
  Life expectancy: Not at all | 4 | 1
  Life expectancy: A little | 5 | 1
  Life expectancy: Moderately | 23 | 2
  Life expectancy: Quite | 38 | 8
  Life expectancy: A lot | 139 | 85
  Life expectancy: Missing | 2 | 0
  Autonomy: Not at all | 2 | 2
  Autonomy: A little | 0 | 1
  Autonomy: Moderately | 7 | 3
  Autonomy: Quite | 23 | 16
  Autonomy: A lot | 178 | 75
  Autonomy: Missing | 1 | 0
  Daily tasks: Not at all | 4 | 0
  Daily tasks: A little | 9 | 1
  Daily tasks: Moderately | 23 | 3
  Daily tasks: Quite | 37 | 19
  Daily tasks: A lot | 136 | 74
  Daily tasks: Missing | 2 | 0
  Social activities: Not at all | 5 | 0
  Social activities: A little | 12 | 0
  Social activities: Moderately | 21 | 4
  Social activities: Quite | 36 | 19
  Social activities: A lot | 135 | 74
  Social activities: Missing | 2 | 0
  Burden of treatment: Not at all | 6 | 6
  Burden of treatment: A little | 6 | 4
  Burden of treatment: Moderately | 25 | 8
  Burden of treatment: Quite | 49 | 24
  Burden of treatment: A lot | 124 | 55
  Burden of treatment: Missing | 1 | 0
  Toxicity: Not at all | 4 | 1
  Toxicity: A little | 4 | 0
  Toxicity: Moderately | 17 | 8
  Toxicity: Quite | 40 | 16
  Toxicity: A lot | 144 | 71
  Toxicity: Missing | 2 | 1
  Economic burden: Not at all | 28 | 17
  Economic burden: A little | 15 | 6
  Economic burden: Moderately | 34 | 13
  Economic burden: Quite | 35 | 16
  Economic burden: A lot | 92 | 45
  Economic burden: Missing | 7 | 0

4. Secondary Outcome: Expectations of Patients 3 Months After Initiation of Treatment
Description: as for outcome 3
Time Frame: 3 months after initiation of treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Number analyzed (Participants) | 155 | 88
Participants
  Treatment efficacy: Not at all | 1 | 0
  Treatment efficacy: A little | 5 | 4
  Treatment efficacy: Moderately | 9 | 5
  Treatment efficacy: Quite | 23 | 10
  Treatment efficacy: A lot | 115 | 68
  Treatment efficacy: Missing | 2 | 1
  Life expectancy: Not at all | 4 | 1
  Life expectancy: A little | 9 | 0
  Life expectancy: Moderately | 18 | 2
  Life expectancy: Quite | 31 | 14
  Life expectancy: A lot | 91 | 70
  Life expectancy: Missing | 2 | 1
  Autonomy: Not at all | 2 | 1
  Autonomy: A little | 2 | 0
  Autonomy: Moderately | 5 | 3
  Autonomy: Quite | 18 | 19
  Autonomy: A lot | 126 | 65
  Autonomy: Missing | 2 | 0
  Daily tasks: Not at all | 2 | 2
  Daily tasks: A little | 11 | 1
  Daily tasks: Moderately | 17 | 4
  Daily tasks: Quite | 38 | 23
  Daily tasks: A lot | 87 | 58
  Daily tasks: Missing | 0 | 0
  Social activities: Not at all | 9 | 1
  Social activities: A little | 14 | 2
  Social activities: Moderately | 20 | 2
  Social activities: Quite | 34 | 22
  Social activities: A lot | 76 | 61
  Social activities: Missing | 2 | 0
  Burden of treatment: Not at all | 16 | 7
  Burden of treatment: A little | 13 | 4
  Burden of treatment: Moderately | 23 | 13
  Burden of treatment: Quite | 41 | 26
  Burden of treatment: A lot | 62 | 38
  Burden of treatment: Missing | 0 | 0
  Toxicity: Not at all | 14 | 2
  Toxicity: A little | 4 | 2
  Toxicity: Moderately | 14 | 8
  Toxicity: Quite | 43 | 25
  Toxicity: A lot | 80 | 51
  Toxicity: Missing | 0 | 0
  Economic burden: Not at all | 31 | 22
  Economic burden: A little | 15 | 1
  Economic burden: Moderately | 10 | 11
  Economic burden: Quite | 30 | 23
  Economic burden: A lot | 67 | 31
  Economic burden: Missing | 2 | 0

5. Secondary Outcome: Stability of Patients in Their Priorities at 3 Months
Description: For each expectation, stability is defined as the prioritization of the expectation at treatment initiation and 3 months after treatment initiation
Time Frame: 3 months after initiation of treatment
Population: Patients without major deviation on study protocol and eligibility criteria who indicated at least one priority in the prioritization grid at the initiation of treatment and 3 months after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Number analyzed (Participants) | 155 | 88
Participants
  Treatment efficacy | 137 | 82
  Life expectancy | 74 | 62
  Autonomy | 119 | 51
  Daily tasks | 59 | 24
  Social activities | 35 | 25
  Burden of treatment | 8 | 1
  Toxicity | 11 | 15
  Economic burden | 2 | 1

6. Secondary Outcome: 1-year Overall Survival
Description: Overall survival is defined as the time between the date of inclusion and the date of death, whatever the cause.
  The rate of overall survival is reported at 1 year
Time Frame: From inclusion to the end of study
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patient
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Number analyzed (Participants) | 211 | 97
percentage of patient | 77.5 [71.4 to 83.0] | 85.2 [76.2 to 90.9]

7. Secondary Outcome: Agreement Rate for Prioritization of Expectations Between Patients and Physicians
Description: For each expectation, the agreement rate is defined by the same prioritization or non-prioritization by the patient-physician pairs.
Time Frame: Day 0 initiation of treatment
Population: Patients without major deviations from study protocol and eligibility criteria who indicated at least one priority in the prioritization grid at treatment initiation and whose physician also indicated at least one priority in the prioritization grid.
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
Number analyzed (Participants) | 200 | 97
Participants
  Treatment efficacy | 174 | 84
  Life expectancy | 123 | 76
  Autonomy | 128 | 47
  Daily tasks | 100 | 45
  Social activities | 122 | 52
  Burden of treatment | 110 | 47
  Toxicity | 91 | 46
  Economic burden | 186 | 93

ADVERSE EVENTS:
Time Frame: 1 year from inclusion.
Description: Only death were assessed on study.
Arm/Group | Elderly Patient (70 Years and Older) | Young Patient (18 Years - 69 Years)
All-Cause Mortality (participants affected / at risk) | 47/211 | 17/97
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT02821793/Prot_SAP_000.pdf